CLINICAL TRIAL: NCT07296848
Title: Health Communications for Adults Smoking Nondaily
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bethany Shorey Fennell (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Bethany Shorey Fennell, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 94633; R03CA286623 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive Health Messaging (PH) (Experimental)
  Interventions: Behavioral: Targeted Smoking Messages
- Negative Health Messaging (NH) (Active Comparator)
  Interventions: Behavioral: Targeted Smoking Messages
- Positive Social Messaging (PS) (Experimental)
  Interventions: Behavioral: Targeted Smoking Messages
- Negative Social Messaging (NS) (Experimental)
  Interventions: Behavioral: Targeted Smoking Messages

INTERVENTIONS:
Behavioral: Targeted Smoking Messages — Participants will view 3 messages within the assigned condition (PH, PS, NH, NS) in a random order. Each message will be displayed for a minimum of 30 seconds.

SUMMARY:
The goal of this study is to develop smoking health risk messaging targeted to adults who smoke some days, but not smoke every day (nondaily). The main purpose is to learn what type of smoking health risk messages will be most likely to encourage adults nondaily to quit completely. Aim 1will iteratively obtain qualitative feedback from adults smoking nondaily on initial message designs, resulting in 12 final messages. Aim 2 will test message properties using a 2 (health vs. social messages) x 2 (positive vs. negative messages) between subjects design to ascertain which messages promote proximal outcomes associated with quitting cigarettes (e.g., new knowledge, risk perceptions, motivation and intentions to quit).

ELIGIBILITY:
Inclusion Criteria:

* individuals that report smoking at least one combustible cigarette per day on 4-28 days in the past 30 days
* able to read/write in English
* able to give informed consent
* no history of daily smoking

Exclusion Criteria:

* enrolled in smoking cessation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge | Baseline and post-intervention (approximately 1 hour)
  Knowledge will be assessed with items based on the ITC-4 (International Tobacco Control (ITC) Four Country Survey) that map onto information presented in the messages (e.g., "Does smoking cause…" heart disease, lung cancer in others; Yes, No, I don't know)
Change in Worry | Baseline and post-intervention (approximately 1 hour)
  Worry will be assessed with 4 items, "How [worried, anxious, fearful, concerned] are you about the effects of smoking?" (1=Not at all, 7=Extremely).
Change in Risk perception | Baseline and post-intervention (approximately 1 hour)
  Risk perceptions will be assessed with 3 items, "If you [don't/do] quit smoking for good, what are your chances of ever developing a smoking-related health problem?" and "How susceptible do you feel you are to developing a smoking-related health problem?" (1=Lowest susceptibility, 7=Highest susceptibility). These will be averaged to form a measure of personal absolute risk
Change in the Contemplation Ladder | Baseline and post-intervention (approximately 1 hour)
  Motivation to quit will be measured with the Contemplation Ladder, rating the position on an 11-rung ladder (0-10) corresponding to stages from "no thought of quitting" (0) to "taking action" (10)
Change in the Motivation to Stop Scale | Baseline and post-intervention (approximately 1 hour)
  Motivation to quit will be measured with the Motivation to Stop Scale, Level of motivation to stop smoking is measured with seven response categories ranging from 1 (lowest) to level 7 (highest level of motivation to stop smoking)
Change in intention to quit | Baseline and post-intervention (approximately 1 hour)
  Intention to quit will be measured with the question "What best describes your intent to stop smoking completely, not even a puff?" (1=Never expect to quit, 4=Will quit in the next 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Shorey Fennell, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No